CLINICAL TRIAL: NCT03960853
Title: Effects of Different Ventilation Modes on Intraoperative Lung Injury and Postoperative Pulmonary Complications in Elderly Patients Undergoing Laparoscopic Colorectal Cancer Resection
Brief Title: Effects of Different Ventilation Patterns on Lung Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Dongxue Li, Principal Investigator, The department of anesthesiology ,Sixth Affiliated Hospital, Sun Yat-sen University, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2019ZSLYEC-184
Record Dates: First submitted 2019-05-19; First posted 2019-05-23 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2019-06

CONDITIONS: Lung Injury
Keywords: aged; mechanical ventilation,
MeSH Terms: conditions — Lung Injury

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pressure-controlled ventilation-volume guaranteed (Experimental): patients will be allocated to pressure-controlled ventilation volume guaranteed in operation
  Interventions: Procedure: pressure-controlled ventilation-volume guaranteed
- volume controlled ventilation (Placebo Comparator): patients will be allocated to volume controlled ventilation in operation
  Interventions: Procedure: volume controlled ventilation

INTERVENTIONS:
Procedure: pressure-controlled ventilation-volume guaranteed — patients will be allocated to pressure-controlled ventilation-volume guaranteed in operation
  Arms: pressure-controlled ventilation-volume guaranteed
Procedure: volume controlled ventilation — patients will be allocated to pressure-controlled ventilation volume guaranteed in operation
  Arms: volume controlled ventilation

SUMMARY:
In 1967, the term "respirator lung" was coined to describe the diffuse alveolar infiltrates and hyaline membranes that were found on postmortem examination of patients who had undergone mechanical ventilation.This mechanical ventilation can aggravate damaged lungs and damage normal lungs. In recent years, Various ventilation strategies have been used to minimize lung injury, including low tide volume, higher PEEPs, recruitment maneuvers and high-frequency oscillatory ventilation. which have been proved to reduce the occurrence of lung injury.

In 2012,Needham et al. proposed a kind of lung protective mechanical ventilation, and their study showed that limited volume and pressure ventilation could significantly improve the 2-year survival rate of patients with acute lung injury.Volume controlled ventilation is the most commonly used method in clinical surgery at present.Volume controlled ventilation(VCV) is a time-cycled, volume targeted ventilation mode, ensures adequate gas exchange. Nevertheless, during VCV, airway pressure is not controlled.Pressure controlled ventilation（PCV） can ensure airway pressure,however minute ventilation is not guaranteed.Pressure controlled ventilation-volume guarantee(PCV-VG) is an innovative mode of ventilation utilizes a decelerating flow and constant pressure. Ventilator parameters are automatically changed with each patient breath to offer the target VT without increasing airway pressures. So PCV-VG has the advantages of both VCV and PCV to preserve the target minute ventilation whilst producing a low incidence of barotrauma pressure-targeted ventilation.

Current studies on PCV-VG mainly focus on thoracic surgery, bariatric surgery and urological surgery, and the research indicators mainly focus on changes in airway pressure and intraoperative oxygenation index.The age of patients undergoing laparoscopic colorectal cancer resection is generally higher, the cardiopulmonary reserve function is decreased, and the influence of intraoperative pneumoperitoneum pressure and low head position increases the incidence of intraoperative and postoperative pulmonary complications.Whether PCV-VG can reduce the incidence of intraoperative lung injury and postoperative pulmonary complications in elderly patients undergoing laparoscopic colorectal cancer resection, and thereby improve postoperative recovery of these patients is still unclear.

DETAILED DESCRIPTION:
One hundred patients undergoing elective laparoscopic colorectal cancer resection (age > 65 years old, body mass index(BMI）18-30 kg/m2, American society of anesthesiologists(ASA )grading Ⅰ - Ⅲ ) will be randomly assigned to volume control ventilation(VCV)group and pressure controlled ventilation-volume guarantee(PCV-VG)group.General anesthesia combined with epidural anesthesia will be used to both groups.

Ventilation settings in both groups are VT 8 mL/kg,inspiratory/expiratory (I/E) ratio 1:2,inspired oxygen concentration (FIO2) 0.5 with air,2.0 L/min of inspiratory fresh gas flow,positive end-expiratory pressure (PEEP) 0 millimeter of mercury （mmHg）,respiratory rate (RR) was adjusted to maintain an end tidal CO2 pressure (ETCO2) of 35 -45 mmHg.

In operation dates will be collected at the following time points: preanesthesia, 1 hour after pneumoperitoneum,2 hours after pneumoperitoneum ,30 minutes after admission to post-anaesthesia care unit (PACU) .The dates collected or calculated are the following:1)peak airway pressure,plate airway pressure, mean inspiratory pressure, dynamic compliance, RR,Exhaled VT andETCO2，2) Arterial blood gas analysis: arterial partial pressure of oxygen (PaO2), arterial partial pressure of carbon dioxide (PaCO2),power of hydrogen（PH）, and oxygen saturation (SaO2)，3) Oxygenation index (OI) calculation; PaO2/FIO2, 4) Ratio of physiologic dead-space over tidal volume(Vd/VT) (expressed in %) was calculated with Bohr's formula ; Vd/VT = (PaCO2 - ETCO2)/PaCO2,5) Hemodynamics: heart rate, mean arterial pressure (MAP),and central venous pressure （CVP），6) lung injury markers ：Interleukin 6(IL6）,Interleukin 8（IL8）,Clara cell protein 16（CC16）,Solution advanced glycation end products receptor（SRAGE）,tumor necrosis factor α(TNFα) .

Investigators will collect the following dates according to following-up after surgery: the incidence of postoperation pulmonary complications(PPC) based on PPC scale within seven days , incidence of pneumonia within seven days after surgery,incidence of atelectasis within seven days after surgery,length of hospital days after surgery, the incidence of postoperative unplanned admission to ICU, the incidence of operation complications within 7 days after surgery, the incidence of postoperative systematic complications within 7 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. scheduled for Laparoscopic colorectal cancer resection
2. age >65 years
3. body mass index(BMI) 18-30kg / m2
4. ASA gradingⅠ-Ⅲ

Exclusion Criteria:

1. history of lung surgery
2. severe restrictive or obstructive pulmonary disease (preoperative lung function test: forced vital capacity(FVC)< 50% predictive value of FVC,forced expiratory volume at one second(FEV1)< 50% predictive value of FEV1
3. Acute respiratory failure, pulmonary infection, ALI/ARDS, and acute stage of asthmaAcute respiratory failure, pulmonary infection, acute lung injury(ALI),acute respiratory distress syndrome(ARDS), and acute stage of asthma (bronchodilators were needed for treatment) were found within 1 month before surgery
4. Patients at risk of preoperative reflux aspiration
5. Preoperative positive pressure ventilation (as obstructive sleep apnea hypopnea syndrome patients) or long-term home oxygen therapy were performed
6. Serious heart, liver and kidney diseases: heart function class more than 3, severe arrhythmia (sinus bradycardia (ventricular rate < 60 times/min), atrial fibrillation, atrial flutter, atrioventricular block, frequent premature ventricular and polyphyly ventricular early, early to R on T, ventricular fibrillation and ventricular flutter), acute coronary syndrome, liver failure, kidney failure
7. Neuromuscular diseases affect respiratory function, such as Parkinson's disease, myasthenia gravis and cerebral infarction affect normal breathing
8. Mental illness, speech impairment, hearing impairment
9. Contraindications for spinal anesthesia puncture
10. Refuse to participate in this study or participate in other studies -

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
occurrence rate of Oxygenation index≤300mmHg | 10minutes before anesthesia,1 hour after pneumoperitoneum,2 hour after pneumoperitoneum,30 minutes after after extubation
  Oxygenation index(OI)=PaO2/FiO2

SECONDARY OUTCOMES:
Occurrence rate of pulmonary complications | Day 0 to 7 after surgery
  Pulmonary complications were assessed using the Postoperation Pulmonary complication ( PPC) scale,The scale is divided into four grades, with 0 indicating no pulmonary complications and 1 to 4 indicating increasingly severe pulmonary complications.
incidence of pneumonia | Day 0 to 7 after surgery
  record the occurrence rate of pneumonia after surgery
incidence of pulmonary atelectasis | Day 0 to 7 after surgery
  record the occurrence rate of pulmonary atelectasis after surgery
peak airway pressure | through mechanical ventilation,average of 3 hours
  Peak airway Pressure（Ppeak, cm H2O)
Plateau airway pressure | through mechanical ventilation,average of 3 hours
  Plateau airway pressure（Pplat, cm H2O）
Static lung compliance | through mechanical ventilation,average of 3 hours
  Static lung compliance (Csta, ml/cm H2O) = Vt/ (Pplat-PEEP)
Dynamic lung compliance | through mechanical ventilation,average of 3 hours
  Dynamic lung compliance (Cdyn , ml/cm H2O)= Vt/ (Ppeak-PEEP)
Arterial partial pressure of oxygen | 10 minutes before anesthesia, 1 hour after pneumoperitoneum, 2 hours after pneumoperitoneum, 30 minutes after extubation
  Arterial partial pressure of oxygen (PaO2, mmHg）
assessing change of Alveolar-arterial oxygen tension difference | 10 minutes before anesthesia, 1 hour after pneumoperitoneum, 2 hours after pneumoperitoneum, 30 minutes after extubation
  Alveolar-arterial oxygen tension difference (mmHg）
assessing change of Respiratory index | 10 minutes before anesthesia, 1 hour after pneumoperitoneum, 2 hours after pneumoperitoneum, 30 minutes after extubation
  Fraction of inspired oxygen (FiO2); Respiratory index (RI) =Ratio of alveolar-arterial oxygen tension difference to FiO2
assessing change of Alveolar dead space fraction | 10 minutes before anesthesia, 1 hour after pneumoperitoneum, 2 hours after pneumoperitoneum,30 minutes after extubation
  Arterial carbon dioxide partial pressure (PaCO2); partial pressure of carbon dioxide in endexpiratory gas (PetCO2); Alveolar dead space fraction (Vd/Vt）=(PaCO2-PetCO2)/ PaCO2;
assessing change of lactic acid | 10 minutes before anesthesia, 1 hour after pneumoperitoneum, 2 hours after pneumoperitoneum, 30 minutes after extubation
  lactate ( LAC), mmol/L
assessing change of Advanced glycation end products receptor | 10 minutes before anesthesia,30 minutes after extubation
  Advanced glycation end products receptor (RAGE, pg/ml)
assessing change of Tumor Necrosis Factor alpha | 10 minutes before anesthesia,30 minutes after extubation
  Tumor Necrosis Factor alpha (TNF-α, pg/ml)
assessing change of Interleukin 6 | 10 minutes before anesthesia,30 minutes after extubation
  Interleukin 6 (IL-6, pg/ml)
assessing change of Interleukin 8 | 10 minutes before anesthesia,30 minutes after extubation
  Interleukin 8 (IL-8, pg/ml)
assessing change of Clara cell protein 16, | 10 minutes before anesthesia,30 minutes after extubation
  Clara cell protein 16,
The occurrence rate of hypoxemia in PACU | 30 minutes after extubation
  The occurrence rate of hypoxemia (SPO2<90% or PaO2<60 mmHg) in PACU
Occurrence rate of operation complications | within 7 days after operation
  abdominal abscess, anastomotic fistula, bleeding and the incidence of reoperation within 7 days
Occurrence rate of Systemic complications | within 7 days after surgery
  Systemic complications including sepsis and septic shock
Antibiotic dosages | within 7 days after surgery
  record the Antibiotic dosages within 7 days after surgery
incidence of Unplanned admission to ICU | within 30 days after surgery
  Unplanned admission to ICU within 30 days after surgery
Length of ICU stay within 30 days after surgery | within 30 days after surgery
  Length of ICU stay within 30 days after surgery
Length of hospital stay within 30 days after surgery | within 30 days after surgery
  Length of hospital stay within 30 days after surgery
Death from any cause | within 30 days after surgery
  Death from any cause 30 days after surgery
The occurrence rate of hypoxemia after surgery | within 7 days after surgery
  The occurrence rate of hypoxemia (SPO2<90% or PaO2<60 mmHg) after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sanqing Jin, MD, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University; Dongxue Li, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Six Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Respirator lung syndrome. Minn Med. 1967 Nov;50(11):1693-705. No abstract available. PMID 5235461
- [Background] Slutsky AS, Ranieri VM. Ventilator-induced lung injury. N Engl J Med. 2013 Nov 28;369(22):2126-36. doi: 10.1056/NEJMra1208707. No abstract available. PMID 24283226
- [Background] Needham DM, Colantuoni E, Mendez-Tellez PA, Dinglas VD, Sevransky JE, Dennison Himmelfarb CR, Desai SV, Shanholtz C, Brower RG, Pronovost PJ. Lung protective mechanical ventilation and two year survival in patients with acute lung injury: prospective cohort study. BMJ. 2012 Apr 5;344:e2124. doi: 10.1136/bmj.e2124. PMID 22491953
- [Background] Ball L, Dameri M, Pelosi P. Modes of mechanical ventilation for the operating room. Best Pract Res Clin Anaesthesiol. 2015 Sep;29(3):285-99. doi: 10.1016/j.bpa.2015.08.003. Epub 2015 Sep 2. PMID 26643095
- [Background] Mahmoud K, Ammar A, Kasemy Z. Comparison Between Pressure-Regulated Volume-Controlled and Volume-Controlled Ventilation on Oxygenation Parameters, Airway Pressures, and Immune Modulation During Thoracic Surgery. J Cardiothorac Vasc Anesth. 2017 Oct;31(5):1760-1766. doi: 10.1053/j.jvca.2017.03.026. Epub 2017 Mar 22. PMID 28673814
- [Background] Dion JM, McKee C, Tobias JD, Sohner P, Herz D, Teich S, Rice J, Barry ND, Michalsky M. Ventilation during laparoscopic-assisted bariatric surgery: volume-controlled, pressure-controlled or volume-guaranteed pressure-regulated modes. Int J Clin Exp Med. 2014 Aug 15;7(8):2242-7. eCollection 2014. PMID 25232415
- [Background] Choi EM, Na S, Choi SH, An J, Rha KH, Oh YJ. Comparison of volume-controlled and pressure-controlled ventilation in steep Trendelenburg position for robot-assisted laparoscopic radical prostatectomy. J Clin Anesth. 2011 May;23(3):183-8. doi: 10.1016/j.jclinane.2010.08.006. Epub 2011 Mar 4. PMID 21377341
- [Background] Tran D, Rajwani K, Berlin DA. Pulmonary effects of aging. Curr Opin Anaesthesiol. 2018 Feb;31(1):19-23. doi: 10.1097/ACO.0000000000000546. PMID 29176377
- [Background] Kalmar AF, Foubert L, Hendrickx JF, Mottrie A, Absalom A, Mortier EP, Struys MM. Influence of steep Trendelenburg position and CO(2) pneumoperitoneum on cardiovascular, cerebrovascular, and respiratory homeostasis during robotic prostatectomy. Br J Anaesth. 2010 Apr;104(4):433-9. doi: 10.1093/bja/aeq018. Epub 2010 Feb 18. PMID 20167583